CLINICAL TRIAL: NCT07231497
Title: Cognitive Strategies in Early Psychosis 1
Acronym: COSTEP 1
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00025500; P50MH119569 (NIH)
Record Dates: First submitted 2025-08-21; First posted 2025-11-17 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Cognition; Healthy Participants
Keywords: Cognition; Decision making; Electroencephalography (EEG); Psychosis
MeSH Terms: conditions — Psychotic Disorders | interventions — Modafinil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- COSTEP 1 (Experimental)
  Interventions: Drug: Modafinil

INTERVENTIONS:
Drug: Modafinil — Single dose of 200mg

SUMMARY:
The goal of this clinical is to learn more about decision making in psychosis spectrum disorders, like schizophrenia. The investigators will ask people who do not have psychosis to take a single dose of modafinil and then complete some brain games on the computer that measure decision making. They hope to improve our understanding of psychosis to help people in the future. The main research questions are:

Does a single dose of modafinil change how people play the brain games? Does a single dose of modafinil change brain activity?

Participants will:

Complete an interview and self-report questionnaires. Complete safety screening activities, like a blood draw, a urine drug test, and an alcohol breathalyzer test.

Take a single dose of modafinil. Complete brain games while wearing an electroencephalography (EEG) cap, before and after taking the single dose of modafinil. EEG measures electrical activity in the brain.

DETAILED DESCRIPTION:
Participants will be asked to complete two appointments in this study. These appointments will ideally be about 1 week apart, but can be up to 1 month apart if needed.

The first appointment is the Intake and Clinical appointment. This visit will take between 30 minutes to 2.5 hours, depending on how many study tasks are needed. Participants in this study may have participated in a sister study, called "State Representation in Early Psychosis 2 (STEP 2)." If so, they will not need to complete many of the intake questionnaires, and it is expected to take about 30 minutes for them to complete this appointment. If they did not participate in STEP 2, participants will need to complete the full intake battery.

During the interview, the investigators will ask questions about a participant's medical and psychiatric history, and current and past mental health symptoms. The investigators will collect demographics, as well as information on the person's social life and quality of life. After the interview, they will complete brain games on their computer.

The second appointment is the EEG + Medication appointment. Participants will come in person to the MHealth Fairview Riverside Campus. The visit will take place in the University of Minnesota Department of Psychiatry. This visit will take about 4-4.5 hours.

First, the investigators will complete safety screening measures. This will include:

* A blood draw for lab testing. They will collect one 3mL tube, which is less than ⅔ of a teaspoon.
* A blood pressure reading.
* A breathalyzer to test for the presence of alcohol.
* A urine drug test to screen for the presence of substances.
* If pregnancy is a physical possibility, a urine pregnancy test will be required.

After screening measures are successfully completed, the investigators will fit an EEG cap onto the participant's head. While this is happening, the participant will complete self-report questionnaires. Once the cap is in place, the participant will play some brain games.

After this, the participant will take a single dose of modafinil. The participant will be provided with a meal while the modafinil metabolizes. Afterwards, they will monitor the participant's vital signs and ask whether they are experiencing any adverse effects.

After the observation period is completed, the participant will complete the same brain games on the computer. The investigators will take another vital signs measurement and ask about adverse effects.

The following day, the investigators will contact the participant via phone to ask whether they experienced any adverse effects after leaving the study appointment. This call should last about 5 minutes.

ELIGIBILITY:
Inclusion Criteria:

* English proficiency, as determined by staff observation and participant self-report
* Estimated IQ at or above 70, as estimated by the cognitive assessments
* Is clinical stable, defined as outpatient status for at least one month prior to study participation
* Has clinically stable doses of medication for at least one month prior to study participation as determined by the PI

  * Participants may have minor adjustments in medication doses in the past 30 days, per PI discretion, but may not have major increases or decreases in dosses, or additions or removal of medications in the past 30 days
  * Participants are to have no changes to medications in the past 7 days before study medication administration (i.e., must have been on a stable dose for at least 7 days prior to receiving the study drug).

Exclusion Criteria:

Medical criteria:

* Presence of the following medical concerns, as determined by the study PI:

  * Major neurological disorder
  * History of head injury with or without prolonged consciousness
  * Any major medical condition that, in the opinion of the PI, would impede participation in the study or would put the participant at additional risk by participating
* History of any of the following as reported by the participant:

  * Renal impairment, injury, or disease
  * Hepatic impairment, injury, or disease
  * Myocardial infarction or heart disease.
* The following cardiac symptoms requiring medical follow-up that, in the opinion of the investigator, would impede participation in the study or would put the participant at additional risk by participating

  * Dsypnea
  * Palpitations
  * Orthopnea
  * Pedal oedema
  * Significant dizziness
  * Syncope
  * Claudication ---Low white blood cell count, or is diagnosed with leukopenia, neutropenia, or agranulocytosis
* Presence of unmanaged hypertension (>140/90) or elevated resting heart rate (>100 bpm)
* Abnormal clinical laboratory values:

  * uACR > 30 mg/g
  * creatinine level >0/95 mg/dL
  * AST or ALT >50 U/L
  * Bilirubin >1.2 mg/dL
  * Total Protein <6 g/dL
* Participant is pregnant, planning to become pregnant, or is breastfeeding
* Participant cannot pass the visual acuity test (e.g., a score lower than 20/25 on the Snellen)
* Takes medications or supplements that have major interactions with modafinil (e.g., ketamine, MAOIs, clomipramine, diazepam, propranolol, warfarin, amphetamine or dextroamphetamine, dexmethylphenidate or methylphenidate)
* Has an allergy to modafinil
* Is currently taking modafinil as a prescription
* Has previously experienced Stevens-Johnson syndrome in response to taking a medication

Mental health criteria:

* Meets criteria for severe substance or alcohol use disorder within 3 months of enrollment
* Lifetime history of stimulant use disorder
* Meets criteria for clinical risk of suicidal behavior, as defined by:

  * Clinician judgment
  * Active suicidal ideation at screening or other appointments
  * Previous intent to act on suicidal ideation with a specific plan and/or preparatory acts within 6 months of enrollment
  * A suicide attempt within 6 months of enrollment
* Meets criteria for a depressive episode within the past month as determined by the diagnostic interview or for a severe or extremely severe depressive episode in the abbreviated battery within the past month
* Meets DSM-5 criteria for, or reports professional diagnosis of, a psychotic, bipolar, or autism spectrum disorder
* Has a family history (1st degree relative) of psychotic, bipolar, or autism spectrum disorder
* Is prescribed psychotropic medications or takes supplements with psychotropic effects (e.g., Nootropics)
* Any other psychiatric symptoms or conditions that, in the opinion of the PI, would impede participation in the study or put the participant at additional risk by participating

Other Criteria:

* Unable or unwilling to provide informed consent
* Unable to demonstrate adequate decisional capacity, in the judgment of the consenting study staff member, to make a choice about participating in the research study
* Participant is illiterate
* Have engaged in significant cognitive training, in the opinion of the PI, in the last year

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 103 (Estimated)
Dates: Start 2025-11-12 (Actual); Primary Completion 2030-04-30 (Estimated); Study Completion 2030-04-30 (Estimated)

PRIMARY OUTCOMES:
Test My Brain - Digit Symbol Coding | Baseline
  A computerized cognitive assessment measuring processing speed. Z scores range from -5 to 5, with a higher score indicating increased cognitive functioning.
Test My Brain - Digit Symbol Coding | Day 7 (EEG + Modafinil Appointment)
  A computerized cognitive assessment measuring processing speed. Z scores range from -5 to 5, with a higher score indicating increased cognitive functioning.
Test My Brain - Verbal Paired Associates Memory | Baseline
  A computerized cognitive assessment measuring verbal memory. Z scores range from -5 to 5, with a higher score indicating increased cognitive functioning.
Test My Brain - Verbal Paired Associates Memory | Day 7 (EEG + Modafinil Appointment)
  A computerized cognitive assessment measuring verbal memory. Z scores range from -5 to 5, with a higher score indicating increased cognitive functioning.
Test My Brain - Matrix Reasoning | Baseline
  A computerized cognitive assessment measuring problem solving. Z scores range from -5 to 5, with a higher score indicating increased cognitive functioning.
Test My Brain - Matrix Reasoning | Day 7 (EEG + Modafinil Appointment)
  A computerized cognitive assessment measuring problem solving. Z scores range from -5 to 5, with a higher score indicating increased cognitive functioning.
Test My Brain - Multiracial Emotion Identification | Baseline
  A computerized cognitive assessment measuring social cognition and emotion recognition skills. Z scores range from -5 to 5, with a higher score indicating increased cognitive functioning.
Test My Brain - Multiracial Emotion Identification | Day 7 (EEG + Modafinil Appointment)
  A computerized cognitive assessment measuring social cognition and emotion recognition skills. Z scores range from -5 to 5, with a higher score indicating increased cognitive functioning.
Electroencaphalography (EEG) - Resting alpha synchrony | Day 7 (EEG + Modafinil Appointment)
  The EEG will measure resting state alpha synchrony in the brain. The primary outcome will be differences in EEG activity before and after modafinil administration.
Electroencaphalography (EEG) - Oscillatory frontal gamma synchrony | Day 7 (EEG + Modafinil Appointment)
  The EEG will measure oscillatory frontal gamma synchrony in the brain. The primary outcome will be differences in EEG activity before and after modafinil administration
Electroencaphalography (EEG) - Task-related reward positivity/P900 | Day 7 (EEG + Modafinil Appointment)
  The EEG will measure task-related reward positivity/P900 activity in the brain. The primary outcome will be differences in EEG activity before and after modafinil administration
Electroencaphalography (EEG) - N1 amplitude | Day 7 (EEG + Modafinil Appointment)
  The EEG will measure N1 amplitude in the brain. The primary outcome will be differences in EEG activity before and after modafinil administration
Dot Pattern Expectancy variation (TOPX) Task - Accuracy | Day 7 (EEG + Modafinil Appointment)
  The TOPX task consists of a series of pattern sequences. One pattern is designated the "A" cue, and another the "X" cue, which requires one response (AX, 60-70% of trials, e.g. respond with the left button), while other sequences require a different response (AY or BX, 12-15% of trials each, or BY, 6-10% of trials, e.g. respond with the right button). Given the strong expectation that X's evokes a valid response, BX trials place demands on the fidelity (stability, memory) of the "B" cue state representation to overcome this tendency. Performance is assessed based on accuracy of responses. The primary outcome will be differences in task accuracy before and after modafinil administration.
Dot Pattern Expectancy variation (TOPX) Task - Response Time | Day 7 (EEG + Modafinil Appointment)
  The TOPX task consists of a series of pattern sequences. One pattern is designated the "A" cue, and another the "X" cue, which requires one response (AX, 60-70% of trials, e.g. respond with the left button), while other sequences require a different response (AY or BX, 12-15% of trials each, or BY, 6-10% of trials, e.g. respond with the right button). Given the strong expectation that X's evokes a valid response, BX trials place demands on the fidelity (stability, memory) of the "B" cue state representation to overcome this tendency. Response time performance is assessed based on the delay in the presentation of the stimuli and the selection of the response. The primary outcome will be differences in response times before and after modafinil administration.
Translational Bandit Task (TBT) - Accuracy | Day 7 (EEG + Modafinil Appointment)
  This is a task variant that uses choice options (neutral images) that are rewarded probabilistically. The rewarded stimulus with the highest reward is changed over time. State learning associated with staying or switching stimuli too quickly (lose-switching) can be evaluated. Performance is assessed based on selection of the option that will yield the highest reward. The primary outcome will be differences in task performance before and after modafinil administration.
Translational Bandit Task (TBT) - Response time | Day 7 (EEG + Modafinil Appointment)
  This is a task variant that uses choice options (neutral images) that are rewarded probabilistically. The rewarded stimulus with the highest reward is changed over time. State learning associated with staying or switching stimuli too quickly (lose-switching) can be evaluated. Performance is assessed based on the delay between the presentation of stimuli and the selection of the response. The primary outcome will be differences in task performance before and after modafinil administration.
Translational Bandit Task (TBT) - Reward Seeking Behavior | Day 7 (EEG + Modafinil Appointment)
  This is a task variant that uses choice options (neutral images) that are rewarded probabilistically. The rewarded stimulus with the highest reward is changed over time. State learning associated with staying or switching stimuli too quickly (lose-switching) can be evaluated. Performance is assessed based on the behavior of reward seeking-whether participants "explore" to find new reward scenarios, or if they stay to "exploit" a known reward scenario. The primary outcome will be differences in reward seeking behavior before and after modafinil administration.

SECONDARY OUTCOMES:
Brief Psychiatric Rating Scale (BPRS) - Global Score | Baseline
  Clinician-administered rating scale to assess psychiatric symptoms such as depression, anxiety, hallucinations, and unusual behavior. Scores on individual items range from 1 (not present) to 7 (extremely severe); global scores range from 24 to 168.

OTHER OUTCOMES:
Abbreviated Quality of Life Scale (aQLS) - Global Score | Baseline
  Clinician-administered rating scale to assess functioning in schizophrenia. Individual items range from 0 (virtually absent) to 6 (Little or no deficit); global scores range from 0 to 54.
Global Functioning - Social Scale (GFS) | Baseline
  Clinician-administered rating scale to assess social functioning. Scores range from 1 (extreme social isolation) to 10 (Superior social/interpersonal functioning).
Global Functioning - Role Scale (GFR) | Baseline
  Clinician-administered rating scale to assess occupational functioning. Scores range from 1 (Extreme role dysfunction) to 10 (Superior role functioning)

CONTACTS AND LOCATIONS:
Overall Officials: Sophia Vinogradov, MD, Principal Investigator — University of Minnesota; Caroline Demro, Ph.D., Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with the NIMH Data Archive (collection ID pending).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be shared 1 year following study completion. There is no end date for data sharing.
Access Criteria: Users who register with the NIMH Data Archive will be able to access the data.